CLINICAL TRIAL: NCT05964582
Title: A Multi-center, Multi-national, Prospective Surveillance Study of Respiratory Syncytial Virus Disease in Infants and Toddlers 6 to < 22 Months of Age
Brief Title: Prospective Surveillance of Respiratory Syncytial Virus Disease in Infants and Toddlers
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: VAD00019; U1111-1281-0204 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-07-07; First posted 2023-07-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy children aged 6 months to < 22 months: No vaccine will be administered. All enrolled participants will have a blood sample collected at enrollment (visit 01) and a nasal swab collected each time they have an RSV-like illness visit

SUMMARY:
The study is a multi-center, multi-national, prospective surveillance study in which the study participants will not receive a study vaccine but will provide a baseline blood sample and be followed for acute respiratory disease during 6 months. The 6-month follow-up will occur for the most part during the Respiratory Syncytial Virus(RSV) season (based on enrollment timing and as per feasibility). A maximum of 1000 children from 6 to < 22 months of age are planned to be enrolled in 5 to 10 countries, 1 to 2 sites per country, targeting approximately 100 participants per country. The purpose of the study is to assess the seroprevalence and incidence of RSV disease during the study period in the targeted countries and sites for a Phase III vaccine study.

DETAILED DESCRIPTION:
The duration of the study will be 6 months for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 months to < 22 months on the day of inclusion (means the day of the 6-month birthday to the day before the 22-month birthday)
* Participants who are healthy as determined by medical evaluation including medical history
* Born at full term of pregnancy (≥ 37 weeks) or born after a gestation period of 27 through 36 weeks and medically stable as assessed by the investigator, based on the following definition: "Medically stable" refers to the condition of premature infants who do not require significant medical support or ongoing management for debilitating disease and who have demonstrated a clinical course of sustained recovery by the time they are enrolled in the study

Exclusion Criteria:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion
* Probable or confirmed ongoing case of viral respiratory infection (including COVID-19, influenza, rhinovirus, etc.) at the time of enrollment. A prospective participant should not be included in the study until the respiratory infection has resolved
* Member of a household that contains an immunocompromised individual, including, but not limited to:

  * a person who is human immunodeficiency virus (HIV) infected
  * a person who has received chemotherapy within the 12 months prior to study enrollment
  * a person who has received (within the past 6 months) or is receiving (at the time of enrollment) immunosuppressant agents
  * a person living with a solid organ or bone marrow transplant
* Participant's mother previous receipt or planned administration of an investigational RSV vaccine during pregnancy and/or breastfeeding
* Receipt or planned receipt of any of the following vaccines:

  * Any intranasal live attenuated vaccine within the 28 days prior to enrollment
  * Any injectable live attenuated vaccine within the 28 days prior to and after enrollment
* Previous receipt of an investigational RSV vaccine or receiving any anti-RSV product (such as ribavirin or RSV immune globulin or RSV monoclonal antibody) less than 6 months before enrollment
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Participation at the time of study enrollment or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial

Ages: 6 Months to 21 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
RSV A serum neutralizing antibody (Nab) titers | At Day 1
  To assess RSV A serum Nab titers overall
RSV A serum neutralizing antibody (Nab) titers | At Day 1
  To assess RSV A serum Nab titers by country
RSV B serum Nab titers | At Day 1
  To assess RSV B serum Nab titers overall
RSV B serum Nab titers | At Day 1
  To assess RSV B serum Nab titers overall by country
Anti-F immunoglobulin A (IgA) and G (IgG) enzyme linked immunosorbant assay (ELISA) titers | At Day 1
  To assess Anti-F IgA and IgG ELISA titers overall
Anti-F immunoglobulin A (IgA) and G (IgG) enzyme linked immunosorbant assay (ELISA) titers | At Day 1
  To assess Anti-F IgA and IgG ELISA titers by country
Baseline serostatus | At Day 1
  To assess baseline serostatus overall
Baseline serostatus | At Day 1
  To assess baseline serostatus by country
Occurrence of ARD associated with any RT PCR confirmed RSV strain during the study | Throughout study, approximately 6 months
  To assess to incidence of ARD confirmed by RT PCR overall
Occurrence of ARD associated with any RT PCR confirmed RSV strain during the study | Throughout study, approximately 6 months
  To assess to incidence of ARD confirmed by RT PCR by country
Occurrence of LRTD associated with any RT PCR confirmed RSV strain during the study | Throughout study, approximately 6 months
  To assess to incidence of LRTD confirmed by RT PCR overall
Occurrence of LRTD associated with any RT PCR confirmed RSV strain during the study | Throughout study, approximately 6 months
  To assess to incidence of LRTD confirmed by RT PCR by country

SECONDARY OUTCOMES:
RSV A serum Nab titers | At Day 1
  To assess RSV A serum Nab titers for each age group overall
RSV A serum Nab titers | At Day 1
  To assess RSV A serum Nab titers for each age group by country
RSV B serum Nab antibody titers | At Day 1
  To assess RSV B serum Nab titers for each age group overall
RSV B serum Nab antibody titers | At Day 1
  To assess RSV B serum Nab titers for each age group by country
Anti-F IgA and IgG ELISA titers | At Day 1
  To assess Anti-F IgA and IgG ELISA titers for each age group overall
Anti-F IgA and IgG ELISA titers | At Day 1
  To assess Anti-F IgA and IgG ELISA titers for each age group by country
Baseline serostatus by age group | At Day 1
  To assess baseline serostatus for each age group overall
Baseline serostatus by age group | At Day 1
  To assess baseline serostatus for each age group by country
Occurrence of ARD associated with any RT PCR confirmed RSV strain during the study | Throughout study, approximately 6 months
  To assess to incidence of ARD confirmed by RT PCR for each age group overall
Occurrence of ARD associated with any RT PCR confirmed RSV strain during the study | Throughout study, approximately 6 months
  To assess to incidence of ARD confirmed by RT PCR for each age group by country
Occurrence of LRTD associated with any RT PCR confirmed RSV strain during the study | Throughout study, approximately 6 months
  To assess to incidence of LRTD confirmed by RT PCR for each age group overall
Occurrence of LRTD associated with any RT PCR confirmed RSV strain during the study | Throughout study, approximately 6 months
  To assess to incidence of LRTD confirmed by RT PCR for each age group by country
Occurrence of ARD associated with each RT-PCR confirmed RSV strain (A/B) during the study | Throughout study, approximately 6 months
  To assess to incidence of ARD confirmed by RT PCR for each strain overall
Occurrence of ARD associated with each RT-PCR confirmed RSV strain (A/B) during the study | Throughout study, approximately 6 months
  To assess to incidence of ARD confirmed by RT PCR for each strain by country
Occurrence of severe LRTD associated with any RT PCR confirmed RSV strain during the study | Throughout study, approximately 6 months
  To assess the severity of LRTD confirmed by any RT PCR for each strain
Occurrence of LRTD associated with each RT-PCR confirmed RSV strain (A/B) during the study | Throughout study, approximately 6 months
  To assess to incidence of LRTD confirmed by RT PCR for each strain overall
Occurrence of LRTD associated with each RT-PCR confirmed RSV strain (A/B) during the study | Throughout study, approximately 6 months
  To assess to incidence of LRTD confirmed by RT PCR for each strain by country
Occurrence of clinically diagnosed RSV ARD according to routine practice (with or without RT-PCR RSV confirmation) during the study | Throughout study, approximately 6 months
Occurrence of clinically diagnosed RSV LRTD according to routine practice (with or without RT-PCR RSV confirmation) during the study | Throughout study, approximately 6 months
Occurrence of AOM episodes during the study | Throughout study, approximately 6 months
Occurrence of ARD and LRTD associated with any RT PCR confirmed RSV strain during the study, RSV A and RSV B serum neutralizing antibody titers, anti-F IgA and IgG ELISA antibody titers | At Day 1
  To assess the association between RT-PCR confirmed RSV ARD and LRTD and RSV A, B, anti-G IgA an IgG ELISA antibodies at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (15):
- United States (2):
  - Quality Clinical Research - 10040 Regency Cir - HyperCore - PPDS Site Number : 8400001, Omaha, Nebraska
  - Senders Pediatrics Site Number : 8400002, Cleveland, Ohio
- Finland (4):
  - Investigational Site Number : 2460002, Helsinki
  - Investigational Site Number : 2460001, Jarvenpaa
  - Investigational Site Number : 2460004, Kokkola
  - Investigational Site Number : 2460003, Tampere
- Ghana (2):
  - Investigational Site Number : 2880002, Kintampo
  - Investigational Site Number : 2880001, Navrongo
- Honduras (2):
  - Investigational Site Number : 3400002, San Pedro Sula
  - Investigational Site Number : 3400001, Tegucigalpa
- India (2):
  - Investigational Site Number : 3560001, Mysuru
  - Investigational Site Number : 3560002, Pune
- Investigational Site Number : 7240001, Móstoles, Madrid, Spain
- Thailand (2):
  - Investigational Site Number : 7640001, Ratchathewi
  - Investigational Site Number : 7640002, Songkhla

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org